CLINICAL TRIAL: NCT01757717
Title: A Pilot Study of Image-Guided Navigation for High Dose Rate Temporary Interstitial Brachytherapy in the Palliative Management of Previously Treated Tumors of the Spine and Pelvis
Brief Title: Image-Guided Navigation for High Dose Rate Temporary Interstitial Brachytherapy in the Palliative Management of Previously Treated Tumors of the Spine and Pelvis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-260
Record Dates: First submitted 2012-12-19; First posted 2012-12-31 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-07

CONDITIONS: Metastatic or Recurrent Lesions in the Spine; Metastatic or Recurrent Lesions in the Pelvis
Keywords: radiation therapy; HDR brachytherapy; Ir-192 high dose rate; 12-260
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Iridium-192

ARMS (1):
- Ir-192 high dose rate (HDR) (Experimental): This pilot study is an investigation into the use of Ir-192 high dose rate (HDR) afterloader-based brachytherapy with catheter placement using image-guided surgical navigation techniques for patients with painful/symptomatic metastatic or recurrent lesions in the spine and/or pelvis that have been maximally treated with external beam radiation therapy.
  Interventions: Radiation: Ir-192 high dose rate (HDR)

INTERVENTIONS:
Radiation: Ir-192 high dose rate (HDR) — Patients will be followed at 2 months (+/- 2 weeks) post-treatment and then approximately every 3 months (+/- 2 weeks) until approximately 11 months of follow up. They will be evaluated for pain referable to the treated site, clinical and radiographic evidence of local progression, and treatment related toxicity. Thereafter, patients will be followed as clinically indicated.

SUMMARY:
The purpose of this study is to see if using a form of imaging during surgery helps the doctors to guide the placement of radiation catheters more accurately.

This method, called "image-guided surgical navigation" may allow the doctors to deliver radiation to the tumor that the patient needs and decrease the amount of radiation delivered to the nearby areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic proof of a malignancy suitable for radiation therapy.
* Patients must have received prior external beam radiation therapy to the region proposed for HDR brachytherapy treatment; evaluation of doses previously delivered to spinal cord/cauda equine, pelvis, and other critical structures (bowel, kidneys, rectum) will be taken into consideration.
* If repeat irradiation would exceed any normal tissue constraint set by MSKCC Radiation Oncology Department dose constraint criteria, the patient will potentially be eligible.
* If the total prior radiation dose to the cord or pelvis exceeds 100 Gy BED equivalent, the patient will be potentially eligible, where a total of 100 BED Gy equivalent is determined by the biological equivalent dose (BED) calculation; BED = nd(1 + d/α/β), where n = number of fractions and d = dose per fraction; α/β is the constant for spinal cord late effect and equals 2. [Rades 2005, Nieder 2005, Sahgal 2012]
* KPS ≥ 60
* Age ≥ 18 years old

Exclusion Criteria:

* Patients who may receive therapeutically effective doses via an external beam approach to the lesion of interest as specified by MSKCC Radiation Oncology Department dose constraint criteria.
* Patients with kyphoplasty cement or hardware that would preclude effective catheter placement.
* Patients with paraspinal extension of disease with visceral involvement.
* Abnormal complete blood count. Any of the following:
* Platelet count < 75,000/ml
* Hb level < 9gm/dl
* WBC < 3.5/ml
* Abnormal coagulation profile: INR > 2.5 and/or PTT > 80
* Patients who are on anticoagulation medication that may not be safely held for the procedure (≥ 5 days for antiplatelet agents and warfarin; ≥ 24 hours for low-molecular weight heparin formulations) will be excluded.
* Contraindications to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ir-192 High Dose Rate (HDR)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ir-192 High Dose Rate (HDR)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 64 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Radiation Dose
Description: Verify feasibility of HDF treatment of spinal and/or pelvic lesions using catheters placed under image-guided navigational techniques, to provide improved dosimetric coverage of lesions such that Cord/Cauda Dmax of <8 Gy
Time Frame: 1 year
Measure: Median (Full Range); unit: cord/cauda max dose in Gy
Arm/Group | Ir-192 High Dose Rate (HDR)
Number analyzed (Participants) | 3
cord/cauda max dose in Gy | 7 [5.8 to 10]

2. Secondary Outcome: Number of Grade 3 of Higher Toxicities
Description: For previously irradiated lesions of the spine and/or pelvis, defined as an acceptable level of severe toxicity (both acute and late effects) in the setting of HDR brachytherapy treatment. Severe toxicity will be defined as ≥ grade 3 NCI CTCAE v 4.0 toxicity that is at least possibly related to treatment
Time Frame: 1 year
Measure: Number; unit: brachytherapy related complications
Arm/Group | Ir-192 High Dose Rate (HDR)
Number analyzed (Participants) | 3
brachytherapy related complications | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ir-192 High Dose Rate (HDR)
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ir-192 High Dose Rate (HDR) (N=3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT01757717/Prot_SAP_000.pdf